CLINICAL TRIAL: NCT03970174
Title: Evaluating the Impact of an Electronic Communication Tool on Patient Experience, ED Visits and Re-hospitalization, and Care Transitions in Hospitalized Patients (Including Those With Dementia): a Mixed Methods Study
Brief Title: Care Transition Patient Experience Study With Electronic Tool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trillium Health Partners (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 828
Record Dates: First submitted 2019-05-09; First posted 2019-05-31 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Care Transition; Communication
Keywords: Patient experience
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: Care Connector care transition module will be rolled out at 2 of 4 wards (intervention) while the other 2 wards will have usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Two of the 4 Medicine wards will have implemented the care transition module of Care Connector
  Interventions: Other: Care Connector care transition module
- Control (No Intervention): Remaining 2 of 4 Medicine wards will use all other aspects of Care Connector (except for care transition module)

INTERVENTIONS:
Other: Care Connector care transition module — Care Connector is an electronic interprofessional communication and collaboration tool. Its features include Physician Sign-Out, documentation, interprofessional care planner, messaging, and flow planner. The newest module is a care transition module which allows physicians to electronically generate discharge summaries as well as incorporation of allied health recommendation, but also will pull information into the PODS (Patient Oriented Discharge Summary) format designed by University Health Network. This results in a patient friendly discharge instruction sheet that can be provided to patient. The intervention arm will have access to the care transition feature, while the control wards do not.
  Arms: Intervention

SUMMARY:
Patients being admitted to hospital are becoming more complex and they often require a team of health professionals (doctors from different disciplines, nurses, and allied health professionals) working together to meet their needs. Effective communication among this team and with patients is essential to providing high quality patient-centered care. Care Connector is an electronic tool that was developed to help health professionals communicate about patient care with each other. It also incorporates best practice whenever possible (such as the used of Patient Oriented Discharge Summary [PODS] developed at University Health Network) during care transitions. We want to understand whether using electronic tools can address the communication issues faced by patients/families, and whether they impact on repeat visits to the Emergency Department or the hospital after discharge. In this study, we will be asking patients and families who have recently been discharged from hospital to describe their experience with communication and care transitions through a brief telephone survey. All of them will be discharged from units where Care Connector was used. However, some of the units would have used the PODS feature while others will not. A small group will also be invited to participate in an in-depth telephone interview. The results of this study will be used to improve Care Connector and to enhance communication and patient experience in general.

DETAILED DESCRIPTION:
In this mixed methods study, we examine how electronic tools impact patient/family experience of communication in hospital and care transitions from hospital to home. Care Connector is an electronic interprofessional communication and collaboration platform initially designed to address communication challenges faced by interprofessional care team. It has been augmented to support care transitions through a care transition module (that include the generation of provider-facing discharge summary and PODS). This study examines the impact of this care transition module on patient/family experience of in-hospital communication and care transitions. The quantitative component is a controlled study where baseline data is collected on 4 medicine wards. The care transition module is then introduced to 2 of the 4 medicine wards (intervention) while the other 2 (control) wards continue to operate without the explicit use of the care transition module. Data is then collected again on all 4 wards to understand impact of patient/family experience, as well as objective outcomes of ED visits and re-admission within 30 days. A number of care transition process measures will also be obtained. In the qualitative component, we will interview patients/families, as well as healthcare providers to understand how technology can or cannot address these issues.

ELIGIBILITY:
Inclusion Criteria:

1. General medical patients cared for and discharged by the Hospitalist service
2. Be 18 years of age and above
3. Length of stay for hospitalization is at least 48 hours
4. The discharge destination is home (with or without support), or retirement home
5. Has the cognitive ability to, or has a substitute decision maker (SDM) (if patient is not capable) able to, provide informed consent for this research study
6. Can be contacted by telephone up to 30 days post discharge
7. Able to respond to survey questions over telephone (assistance from family member or other caregiver at the time of telephone survey is permitted)

Exclusion Criteria:

1. Discharged from a non-Medicine ward (e.g. medicine patient bed spaced to a surgical ward) or from the Emergency Department directly
2. Previously participated in this study (in case of re-admission)
3. Discharge destination is another acute care facility, rehab, palliative care unit, complex continuing care, long term care, or any other facility not listed in inclusion criteria 4.
4. Died in hospital
5. Unable to give informed consent due to language barrier and lack of suitable assistance from family members and/or caregivers and/or SDM (if patient is not capable)
6. Cannot be contacted by telephone after discharge
7. Unable to respond to telephone survey questions for any reason (e.g. hearing impairment, language barrier) and lack of availability of family members and/or other caregivers willing and able to provide assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Care transition measure 3 | Up to 30 days post discharge
  This is a validated measure developed by Coleman et al (Med Care. 2008 Mar;46(3):317-22) to measure quality of care transitions. It contains 3 questions (please see reference for questions).

SECONDARY OUTCOMES:
In-hospital communication | Up to 30 days post discharge
  Subset of questions from the Canadian Patient Experience Survey - Inpatient Care (CPES-IC)
ED visit | 30 days post discharge
  ED visit to any site at Trillium Health Partners
Hospitalization | 30 days post discharge
  Hospitalization to any site at Trillium Health Partners
Presence of follow up plan in discharge summary | At the time of patient discharge (0 days)
  Binary (yes/no) assessment of whether the dictated discharge summary contains a follow-up plan section.
Proportion of appointments with date/time confirmed at discharge | At time of patient discharge (0 days)
  Number of appoints with date/time confirmed / total number of appointments
Proportion of patients referred to community support services | At time of patient discharge (0 days)
  Number of patients referred to community support services / total number of patients

OTHER OUTCOMES:
Subgroup analysis of patients with dementia | Up to 30 days post patient discharge
  We will determine whether a patient has dementia by reviewing all dictated consultation notes and discharge summaries in the medical record to look for mention of dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Tang, MD, Principal Investigator — Trillium Health Partners
Locations (1):
- Trillium Health Partners, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahn-Goldberg S, Okrainec K, Huynh T, Zahr N, Abrams H. Co-creating patient-oriented discharge instructions with patients, caregivers, and healthcare providers. J Hosp Med. 2015 Dec;10(12):804-7. doi: 10.1002/jhm.2444. Epub 2015 Sep 25. PMID 26406116
- [Background] Parry C, Mahoney E, Chalmers SA, Coleman EA. Assessing the quality of transitional care: further applications of the care transitions measure. Med Care. 2008 Mar;46(3):317-22. doi: 10.1097/MLR.0b013e3181589bdc. PMID 18388847
- [Background] Tang T, Lim ME, Mansfield E, McLachlan A, Quan SD. Clinician user involvement in the real world: Designing an electronic tool to improve interprofessional communication and collaboration in a hospital setting. Int J Med Inform. 2018 Feb;110:90-97. doi: 10.1016/j.ijmedinf.2017.11.011. Epub 2017 Nov 22. PMID 29331258
- See also: Canadian Patient Experiences Survey - Inpatient Care (Canadian Institute for Health Information) — https://www.cihi.ca/en/health-system-performance/quality-of-care-and-outcomes/patient-experience